CLINICAL TRIAL: NCT02359565
Title: A Safety and Preliminary Efficacy Trial of Pembrolizumab (MK-3475) in Children With Recurrent, Progressive or Refractory Diffuse Intrinsic Pontine Glioma (DIPG), Non-Brainstem High-Grade Gliomas (NB-HGG), Ependymoma, Medulloblastoma or Hypermutated Brain Tumors
Brief Title: Pembrolizumab in Treating Younger Patients With Recurrent, Progressive, or Refractory High-Grade Gliomas, Diffuse Intrinsic Pontine Gliomas, Hypermutated Brain Tumors, Ependymoma or Medulloblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00130; NCI-2015-00130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-045; PBTC-045 (Other: Pediatric Brain Tumor Consortium); PBTC-045 (Other: CTEP); UM1CA081457 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-02-10 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Constitutional Mismatch Repair Deficiency Syndrome; Lynch Syndrome; Malignant Glioma; Recurrent Brain Neoplasm; Recurrent Childhood Ependymoma; Recurrent Diffuse Intrinsic Pontine Glioma; Recurrent Medulloblastoma; Refractory Brain Neoplasm; Refractory Diffuse Intrinsic Pontine Glioma; Refractory Ependymoma; Refractory Medulloblastoma
MeSH Terms: conditions — Turcot syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Glioma; Brain Neoplasms; Familial ependymoma; Diffuse Intrinsic Pontine Glioma; Medulloblastoma; Ependymoma | interventions — Specimen Handling; Diffusion Tensor Imaging; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 34 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo standard MRI, DCE permeability MRI, DTI, DSC perfusion MRI, MR diffusion imaging and may undergo MR spectroscopy as well as CSF and blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Conventional Magnetic Resonance Imaging; Procedure: Diffusion Tensor Imaging; Procedure: Diffusion Weighted Imaging; Procedure: Dynamic Contrast-enhanced MR Perfusion; Procedure: Dynamic Susceptibility Contrast-Perfusion-Weighted Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Conventional Magnetic Resonance Imaging — Undergo standard MRI
  Other Names: Conventional MRI
Procedure: Diffusion Tensor Imaging — Undergo DTI
  Other Names: DIFFUSION TENSOR MRI; DT-MRI; DTI
Procedure: Diffusion Weighted Imaging — Undergo MR diffusion imaging
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DW-MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Procedure: Dynamic Contrast-enhanced MR Perfusion — Undergo DCE permeability MRI
  Other Names: DCE; DCE MR Perfusion; Dynamic Contrast-enhanced Magnetic Resonance Imaging Perfusion; Dynamic Contrast-enhanced MRI Perfusion; Permeability MRI
Procedure: Dynamic Susceptibility Contrast-Perfusion-Weighted Imaging — Undergo DSC perfusion MRI
  Other Names: DSC; DSC-PWI; Dynamic Susceptibility Contrast Perfusion Weighted Imaging; Dynamic Susceptibility Contrast Perfusion-Weighted MR Imaging; Dynamic Susceptibility Contrast-Enhanced MR Perfusion
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MR spectroscopy
  Other Names: Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; MS
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase I trial studies the side effects and best dose of pembrolizumab and to see how well it works in treating younger patients with high-grade gliomas (brain tumors that are generally expected to be fast growing and aggressive), diffuse intrinsic pontine gliomas (brain stem tumors), brain tumors with a high number of genetic mutations, ependymoma or medulloblastoma that have come back (recurrent), progressed, or have not responded to previous treatment (refractory). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may induce changes in the body's immune system, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety and describe adverse effects associated with administration of the adult recommended dose of pembrolizumab (MK-3475) in each stratum separately.

II. To estimate the sustained objective response rate, (complete response [CR] + partial response [PR], sustained for at least 9 weeks) associated with pembrolizumab (MK-3475) treatment for pediatric patients with recurrent, progressive or refractory diffuse intrinsic pontine glioma (DIPG), non-brainstem high grade glioma (NB-HGG), ependymoma or medulloblastoma.

III. To establish the safety and describe adverse effects associated with administration of the adult recommended dose of pembrolizumab (MK-3475) in pediatric patients with progressive or recurrent hypermutated tumors, including those with constitutional mismatch-repair deficiency (CMMRD) syndrome.

IV. To estimate the sustained response rate of pediatric patients with progressive or recurrent hypermutated NB-HGG, including those with CMMRD syndrome, treated with pembrolizumab (MK-3475).

V. To determine changes in the immunophenotypic profile of PD-1hi CD8+ T cells from serial peripheral blood samples obtained before and during treatment with pembrolizumab (MK-3475) in pediatric patients with hypermutated brain tumors, including those with CMMRD syndrome.

SECONDARY OBJECTIVES:

I. To assess the relationship between outcome (response and progression-free survival) and potential biomarkers, including PD-L1 expression, patient immunophenotype, ribonucleic acid (RNA) signature profile, mutational profile, tumor gene expression and circulating tumor deoxyribonucleic acid (DNA) (ctDNA).

II. To estimate the duration of objective response in patients with measurable disease at baseline and estimate progression-free/event-free/overall survival for patients in each stratum treated with pembrolizumab (MK-3475).

III. To evaluate PD-L1 expression on archival tissue obtained from pediatric patients with eligible primary central nervous system (CNS) tumors.

IV. To examine the ability of quantitative magnetic resonance (MR) spectroscopy and diffusion/weighted imaging/apparent diffusion coefficient (ADC) mapping to provide early assessment of tumor behavior and specifically distinguish pseudoprogression/tumor inflammation from tumor progression.

V. To explore the use of serial MR permeability (dynamic contrast-enhanced [DCE]) and MR perfusion (dynamic susceptibility contrast [DSC]) to determine if elevated relative cerebral blood volume (rCBV) and transfer coefficient (ktrans) can distinguish pseudoprogression/tumor inflammation from tumor progression in tumors treated on this protocol.

VI. To characterize biomarkers, patient immunophenotyping, mutational load (as determined by whole exome sequencing), the tumor gene expression profile and ctDNA in patients receiving pembrolizumab (MK-3475).

VII. To estimate the duration of objective response, progression-free survival/event free survival and document overall survival of pediatric patients with progressive or recurrent hypermutated NB-HGG, including those with CMMRD syndrome, treated with pembrolizumab (MK-3475).

VIII. To estimate the progression-free survival (PFS) of all patients enrolled on stratum C and sustained objective response rate of pediatric patients with hypermutated progressive low grade gliomas including those with CMMRD, treated with pembrolizumab (MK-3475).

IX. To categorize the T-cell receptor repertoire in PD-1+ cells obtained from peripheral blood or from tumor tissue, when available, before and after treatment with pembrolizumab (MK-3475) in pediatric patients treated in stratum C (hypermutated brain tumors).

X. To define the specificity of T-cell receptors against tumor antigens identified in objective IX.

XI. To characterize functional features of T-cell populations after pembrolizumab (MK-3475) treatment and relate these findings to epigenetic programs within these cells.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 34 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo standard magnetic resonance imaging (MRI), dynamic contrast-enhanced magnetic resonance (MR) perfusion (DCE permeability) MRI, diffusion tensor imaging (DTI), dynamic susceptibility contrast-perfusion-weighted imaging (DSC perfusion) MRI, diffusion weighted imaging (MR diffusion imaging) and may undergo MR spectroscopy as well as cerebrospinal fluid (CSF) and blood sample collection during screening and on study.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR STRATA A, B, D AND E
* Tumor: patient must have one of the following diagnoses to be eligible:
* Stratum A, currently closed to enrollment: Patients must have a recurrent, progressive or refractory DIPG following radiation therapy with or without chemotherapy

  * Histologic diagnosis is not required for patients with typical imaging findings of DIPG (defined as patients with a diffuse expansile mass centered in and involving at least 2/3 of the pons); patients with brainstem tumors who have undergone biopsy with a diagnosis of high-grade glioma or diffuse infiltrating glioma are also eligible
* Stratum B: Patients must have a histologically confirmed diagnosis of a non-brainstem high-grade glioma (NB-HGG) that is recurrent, progressive or refractory following therapy which included radiotherapy; spinal primary disease is eligible
* Stratum D: Patients must have a histologically confirmed diagnosis of ependymoma that is recurrent, progressive or refractory following therapy which included radiotherapy
* Stratum E: Patients must have a histologically confirmed diagnosis of medulloblastoma that is recurrent, progressive or refractory following therapy which included radiotherapy
* Patients must have adequate pre-trial formalin-fixed paraffin-embedded (FFPE) tumor material available for use in the biology studies mutational analysis and genome wide sequencing for each stratum

  * Patients with DIPG who have tissue available are requested to submit similar tissue as patients in other strata; however, this is not required for eligibility
* All subjects must have measurable disease in 2-dimensions on MRI scan of the brain; disease should be consistently measured with the two largest perpendicular dimensions
* Patient must be >= 1 but =< 18 years of age at the time of enrollment during the safety portion. Patients < 22 may be enrolled during the efficacy portion of the study.
* Patients must have received prior radiation therapy and/or chemotherapy and recovered from the acute treatment related toxicities (defined as =< grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study; there is no upper limit to the number of prior therapies that is allowed
* Patients must have received their last dose of known myelosuppressive anticancer therapy at least three (3) weeks prior to study enrollment or at least six (6) weeks if prior nitrosourea
* Biologic or investigational agent (anti-neoplastic): Patient must have received their last dose of the investigational or biologic agent >= 7 days prior to study enrollment

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration must be discussed with and approved by the study chair
* Monoclonal antibody treatment and/or agents with prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent >= 28 days prior to study enrollment
* Patient must have completed immunotherapy (e.g. tumor vaccines, oncolytic viruses, etc.) at least 42 days prior to enrollment
* Patients must have had their last fraction of:

  * Craniospinal irradiation >= 3 months prior to enrollment
  * Other substantial bone marrow irradiation >= 6 weeks prior to enrollment
  * Local palliative radiation therapy (XRT) (small port) >= 2 weeks
* Patient must be >= 12 weeks since autologous bone marrow/stem cell transplant prior to enrollment
* Patients must be fully recovered from all acute effects of prior surgical intervention
* Both males and females of all races and ethnic groups are eligible for this study
* Patients with neurological deficits should have deficits that are completely stable for a minimum of 1 week (7 days) prior to enrollment
* Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within two weeks of enrollment must be >= 70; patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Absolute neutrophil count >= 1000 cells/uL
* Platelets >= 75,000 cells /uL (unsupported, defined as no platelet transfusion within 7 days)
* Hemoglobin >= 8 g/dl (may receive transfusions)
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Albumin >= 2 g/dl
* Serum creatinine based on age/gender as noted below; patients that do not meet the criteria below but have a 24 hour creatinine clearance or glomerular filtration rate (GFR) (radioisotope or iothalamate) >= 70 ml/min/1.73 m^2 are eligible

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male); 0.6 (female)
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male); 0.8 (female)
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male); 1 (female)
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* Pulse oximetry > 93% on room air and no evidence of dyspnea at rest
* Human immunodeficiency virus (HIV)- infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients must be off all colony-forming growth factor(s) for at least 1 week prior to registration (e.g. filgrastim, sargramostim, erythropoietin); 2 weeks must have elapsed for long-acting formulations
* Patients must be willing to use brief courses (at least 72 hours) of steroids as directed for potential inflammatory side effects of the therapy if recommended by their treating physician
* Female subjects of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; pregnant women are excluded from this study because pembrolizumab (MK-3475) is an agent with the potential for teratogenic effects; because there is unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab (MK-3475), breastfeeding should be discontinued if the mother is to be treated with pembrolizumab (MK-3475)
* Patients of childbearing or child fathering potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity while being treated on this study and for 4 months after the last dose of study medication
* The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document, inclusive of assent where appropriate, according to institutional guidelines
* STRATUM C: Diagnosis of hypermutated brain tumors Patients with brain tumors and increased tumor mutation burden as determined by

  * Confirmed diagnosis of CMMRD syndrome by Clinical Laboratory Improvement Act (CLIA)-certified germline gene sequencing OR
  * Confirmation of high mutation burden by whole genome/exome sequencing performed in a CLIA-certified laboratory and/or the use of Foundation One next generation sequence panel or another CLIA approved targeted sequencing lab with publicly available correlations between number of mutations found in the panel and mutations per megabase and/or genome; for protocol purposes a high mutation burden will be defined as at least 180 non-synonymous coding-region mutations by whole exome/genome sequencing (well above two standard deviations of the number of median similar mutations described in pediatric CNS cancers) AND/OR a high tumor mutation burden (TMB) or intermediate TMB based on the reporting parameters of the panel; TMB parameters provided for the Foundation One panel are as follows: high TMB is >= 20 mutations per megabase or intermediate TMB is between 6 to 19 mutations per megabase OR
  * Confirmed diagnosis of Lynch syndrome by CLIA-certified germline gene sequencing; patients with Lynch syndrome will not be accounted for in primary objective unless their tumors are determined to have the minimum number of mutations described above but they will still be eligible for this study

    * Low-grade tumors in patients with CMMRD or Lynch syndrome do not have to reach the threshold of 100 mutations for study inclusion
* STRATUM C: Patients must have a histologically confirmed primary brain tumor that is recurrent, progressive or refractory; inclusion criteria encompasses all types of brain tumors (e.g. gliomas, embryonal tumors or any other type of brain tumor as long as other eligibility criteria are met;

  * Patients with high-grade gliomas are eligible for this clinical trial at least 2 weeks after completion of radiotherapy independent of tumor progression/recurrence as long as they are not enrolled on any other therapeutic clinical trial and there is macroscopic residual disease
  * Patients with other concomitant tumors associated with CMMRD and Lynch syndrome including gastrointestinal polyps/adenomas and carcinomas, lymphomas and leukemias will be eligible as long as they are not requiring anticancer therapy directed against these other cancers and meet all other eligibility criteria
* STRATUM C: Patients must have adequate pre-trial FFPE tumor material available and be willing to provide a blood sample for use in the genome wide sequencing studies; while tissue is required for genome-wide sequencing of tumor and germline samples, patients will be deemed eligible for the study with a minimum of approximately 10 unstained slides for the planned analysis
* STRATUM C: Subjects must have measurable disease in 2-dimensions on MRI scan of the brain and/or spine with the exception allowed for non-progressed HGGs; disease should be consistently measured with the two largest perpendicular dimensions
* STRATUM C: Patient should be < 30 years at the time of enrollment
* STRATUM C: Patients must have received prior radiotherapy and/or chemotherapy with the following exceptions:

  * Patients with secondary CNS cancers after a previous medical problem/malignancy who cannot receive full dose of radiotherapy (> 50 Gy) as long as they meet all other eligibility criteria
  * Patients with progressive low-grade gliomas and CMMRD or Lynch syndrome Patients must have recovered from the acute treatment related toxicities (defined as =< grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study; there is no upper limit to the number of prior therapies that is allowed
* STRATUM C: Patients must have received their last dose of known myelosuppressive anticancer therapy at least three (3) weeks prior to study enrollment or at least six (6) weeks if prior nitrosourea
* STRATUM C: Patient must have received their last dose of the investigational or biologic agent >= 7 days prior to study enrollment

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration must be discussed with and approved by the study chair
* STRATUM C: Monoclonal antibody treatment and/or agents with prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent >= 28 days prior to study enrollment
* STRATUM C: Patient must have completed immunotherapy (e.g. tumor vaccines, oncolytic viruses, etc.) at least 42 days prior to enrollment
* STRATUM C: Patients must have had their last fraction of:

  * Craniospinal irradiation >= 3 months prior to enrollment
  * Other substantial bone marrow irradiation >= 6 weeks prior to enrollment
  * Local palliative XRT (small port) >= 2 weeks
* STRATUM C: Patient must be:

  * >= 12 weeks since autologous bone marrow/stem cell transplant prior to enrollment
  * >= 5 years since allogeneic stem cell transplant prior to enrollment with no evidence of active graft versus (vs.) host disease
* STRATUM C: Patients must be fully recovered from all acute effects of prior surgical intervention
* STRATUM C: Both males and females of all races and ethnic groups are eligible for this study
* STRATUM C: Patients with neurological deficits should have deficits that are completely stable for a minimum of 1 week (7 days) prior to enrollment
* STRATUM C: Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within two weeks of enrollment must be >= 60; patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* STRATUM C: Absolute neutrophil count >= 1000 cells/uL
* STRATUM C: Platelets >= 75,000 cells/uL (unsupported, defined as no platelet transfusion within 7 days)
* STRATUM C: Hemoglobin >= 8 g/dl (may receive transfusions)
* STRATUM C: Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* STRATUM C: ALT (SGPT) =< 3 x institutional upper limit of normal
* STRATUM C: Albumin >= 2 g/dl
* STRATUM C: Serum creatinine based on age/gender as noted below; patients that do not meet the criteria below but have a 24 hour creatinine clearance or GFR (radioisotope or iothalamate) >= 70 ml/min/1.73 m^2 are eligible

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male); 0.6 (female)
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male); 0.8 (female)
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male); 1 (female)
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* STRATUM C: Pulse oximetry > 93% on room air and no evidence of dyspnea at rest
* STRATUM C: HIV- infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* STRATUM C: Patients must be off all colony-forming growth factor(s) for at least 1 week prior to registration (i.e. filgrastim; sargramostim; erythropoietin); 2 weeks must have elapsed for long-acting formulations
* STRATUM C: Patients must be willing to use brief courses (at least 72 hours) of steroids as directed for potential inflammatory side effects of the therapy if recommended by their treating physician
* STRATUM C: Female subjects of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; pregnant women are excluded from this study because pembrolizumab (MK-3475) is an agent with the potential for teratogenic effects; because there is unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab (MK-3475), breastfeeding should be discontinued if the mother is to be treated with pembrolizumab (MK-3475)
* STRATUM C: Patients of childbearing or child fathering potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity while being treated on this study and for 4 months after the last dose of study medication
* STRATUM C: The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document, inclusive of assent where appropriate, according to institutional guidelines

Exclusion Criteria:

* EXCLUSION CRITERIA FOR STRATA A, B, D AND E
* Concurrent Illness

  * Patients with active autoimmune disease or documented history of autoimmune disease/syndrome that requires ongoing systemic steroids or systemic immunosuppressive agents, except

    * Patients with vitiligo or resolved asthma/atopy
    * Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome
  * History of or ongoing pneumonitis or significant interstitial lung disease Note: This would include non-infectious pneumonitis that required steroid use
  * Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results
  * Patients with other current malignancies
  * Patients with known hypermutated brain tumors including those with CMMRD and Lynch syndrome are ineligible for enrollment in Strata A, B, D and E
  * Patients who have received a solid organ transplant
* Patients with bulky tumor on imaging are ineligible; treating physicians are encouraged to contact the study chair to request a rapid central imaging review to confirm fulfilment of these eligibility criteria, if they have concerns

Bulk tumor is defined as:

* Tumor with evidence of clinically significant uncal herniation or midline shift
* Tumor with diameter of > 5 cm in one dimension on T2/fluid attenuated inversion recovery (FLAIR)
* Tumor that in the opinion of the site investigator, shows significant mass effect in either the brain or spine
* Multi-focal/ metastatic disease:

Note: Multiple foci of enhancement in a single FLAIR abnormality is permissible and will not exclude the subject

* Patients with multi-focal parenchymal disease are ineligible
* Patients with leptomeningeal metastatic disease are eligible; this includes disease that is discrete from the primary lesion but that has a radiographic appearance consistent with leptomeningeal spread, rather than likely trans-parenchymal spread

  * Strata B, D and E - patients whose tumor has a significant component involving the brainstem or with significant fourth ventricular compression are ineligible

    * Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible
    * Patients who have a known active hepatitis B or hepatitis C infection are ineligible; patient must have documented evidence of negative tests for the presence of hepatitis B surface antigen and hepatitis C (anti-hepatitis C virus [HCV] antibody OR hepatitis [Hep] C RNA-qualitative)
    * Patients who have received the last vaccination of a live vaccine =< 30 days prior to enrollment are ineligible; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist [registered trademark]) are live attenuated vaccines, and must meet timeline for live vaccine
    * Patients with a history severe (>= grade 3) hypersensitivity reaction to a monoclonal antibody are ineligible
    * Patients who have received previous therapy with an anti-CTLA4, anti-CD137

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Within 30 days of treatment
  Will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All adverse events observed during the dose finding period as well as during later courses will be summarized by stratum and by dose (if applicable). Separate tables for adverse events attributable to pembrolizumab will also be provided for each of the five strata.
Sustained objective response (partial response + complete response) | Within 12 cycles (approximately 9 months)
  Stratum specific exact confidence interval estimates will be provided for the sustained objective response rates. In addition, if adequate number of responses is observed to make such analyses meaningful, stratum-specific confirmed sustained objective response rates observed during treatment will be estimated by cumulative incidence functions.
Change in the percentage of CD8+ T cells that are PD-1+ due to treatment with pembrolizumab (Stratum C) | Baseline to after 6 weeks of treatment
  A 1-sample t-distribution-based confidence interval (or its non-parametric counterparts, as needed) will be used to estimate the average change in the percentage of CD8+ T cells that are PD-1+ due to treatment with pembrolizumab.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Date of initial treatment to the earliest date of disease progression or death from any cause for patients who fail and to the date of last contact for patients who remain at risk for failure, assessed bi-annually up to 3 years and then yearly thereafter
  Log-ranks tests or Cox regression models will be used to explore associations between biomarkers and PFS and OS.
Event-free survival | Up to 3 years
  Kaplan-Meier estimates of event free survival distribution for all evaluable patients within each stratum will be provided.
Overall survival (OS) | Date of diagnosis to the earliest date of death from any cause or to the date of last contact for patients who remain at risk for failure, assessed bi-annually up to 3 years and then yearly thereafter
  Kaplan-Meier estimates of OS distribution for all evaluable patients within each stratum will be provided. Log-ranks tests or Cox regression models will be used to explore associations between biomarkers and progression free survival (PFS) and OS.
Radiologic response (Stratum C) | Up to 3 years
  Will report any objective radiological responses observed in subjects who were not part of the primary cohort of progressive/recurrent high-grade gliomas (HGGs).
Biomarker expression levels | Up to 18 cycles (approximately 13.5 months)
  The biomarker data generated as part of this study will be summarized via descriptive statistics and plots. The association between response and potential biomarkers will be evaluated by Fisher's exact or Chi-square test for categorical outcomes and two sample t-tests (or appropriate non-parametric counterparts) for continuous outcomes. Log-ranks tests or Cox regression models will also be used to explore associations between biomarkers and PFS and OS. These analyses will be done in a stratum specific fashion.
Changes in quantitative imaging parameters | Baseline to up to 34 cycles (approximately 25.5 months)
  Observed values of the proposed quantitative imaging parameters as well as changes in these parameters across time will be described and summarized via descriptive statistics and plots. Mixed effects models will be used to explore differences in estimated slope parameters of the quantitative imaging. Pairwise changes in these imaging parameters across various time points will also be described. T-tests (or their non-parametric equivalent) will be used to compare differences in pairwise changes between patients with progression vs. pseudoprogression/tumor inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene I Hwang, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (12):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada